CLINICAL TRIAL: NCT04840797
Title: HeartStart HS1 Defibrillator* Event Registry
Status: Recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: TC_ECR_HS1_2020_10819
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Sudden Cardiac Arrest
Keywords: AED; Post -Market; Cardiology
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Suspected Sudden Cardiac Arrest: All subjects with suspected of a circulatory arrest of any cause.
  Interventions: Device: HeartStart HS1

INTERVENTIONS:
Device: HeartStart HS1 — Automated External Defibrillator

SUMMARY:
A Prospective study on the performance and safety of the HeartStart OnSite (Model M5066A) & HeartStart Home (Model M5068A) Defibrillator device data.

DETAILED DESCRIPTION:
The objective of this PMCF (Post Market Clinical Follow-up) prospective collection of post-event data registry is to confirm the safety and performance as expressed in the energy delivery by the HeartStart HS1 Defibrillator (HeartStart OnSite and Home models in North America) in the population for the device's intended use in reference to its commercial labeling, and in relationship to the type of pads attached to the device.

ELIGIBILITY:
Inclusion Criteria:

* Have been suspected of a circulatory arrest for any cause.
* Have had HeartStart HS1 Defibrillator with electrodes:

Adult SMART Pads Cartridge [REF: M5071A], Infant/Child SMART Pads Cartridge (REF:M5072A) applied to their body and powered up with HS1 battery (Model M5070A), regardless of whether a defibrillation shock was delivered

Exclusion Criteria:

* Subjects will be excluded if any of the following are present:
* AED or pad use other than the HeartStart HS1 Defibrillator with above referenced Philips electrode pads. Note: Use of a device other than the Philips HeartStart HS1 AED does not preclude enrollment if the AED or an Advanced Life Support defibrillator was used after the HeartStart HS1 AED.
* AED used for training purposes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone who is suspected of having a sudden cardiac arrest.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean shock energy delivered in the pediatric population | Up to 15 minutes during device placement
  Mean of shock energy delivered, when the pediatric defibrillation pads were attached to the AED as intended for infants and children under 25 kilograms / 55 pounds or 0-8 years old.
Mean shock energy delivered in the adult population | Up to 15 minutes during device placement
  Mean of shock energy delivered, when the adult defibrillation pads were attached to the AED as intended for in children and adults over 25 kilograms / 55 pounds or greater than 8 years old.
The Patient Analysis System (PAS) shock advisory algorithm performance as determined by evaluation of the ECG as aligned with the device advisement. | Up to 15 minutes during device placement
  Performance is defined by the sensitivity and specificity; positive predictive value and false positive rate will be reported for each rhythm category (as defined by device labeling).
Accurate detection of shockable rhythms and facilitation of shocks. | Up to 15 minutes during device placement
  The percentage of events where a shockable rhythm was identified by the device, the device advised a shock, and the device delivered a shock when the shock button was pressed.
Defibrillation success | Up to 15 minutes during device placement
  Defibrillation success and the number of shocks required for success.

SECONDARY OUTCOMES:
Frequency and severity of unexpected adverse events | Up to 15 minutes during device placement
  Frequency and severity of unexpected adverse events
Unanticipated adverse device effects (UADE) | Up to 15 minutes during device placement
  Unanticipated adverse device effects (UADE)
Median operating time intervals | Up to 15 minutes during device placement
  Median operating time intervals
Routine self-test performance/Battery Insertion self-test performance | Up to 15 minutes during device placement
  Routine self-test performance/Battery Insertion self-test performance
Device arming after shock advisement. | Up to 15 minutes during device placement
  The percentage of events where the device advised a shock and the device armed.
Energy delivered consistent with device labeling | Up to 15 minutes during device placement
  The percentage of defibrillations in which the energy delivered was consistent with device labeling.
Pad replacement notification | Up to 15 minutes during device placement
  Number of events in which pads were replaced at any time during the event after the user is prompted to do so by the device
Shock button effectively pressed after shock advisement | Up to 15 minutes during device placement
  The percentage of events where a shock was recommended by the device and the shock button was pressed.
Indicators of battery status/depletion (device logged data) | Up to 15 minutes during device placement
  Percentage of events that include indicators of battery status/depletion (device logged data)
Aborted shocks because of low or high impedance | Up to 15 minutes during device placement
  Percentage of aborted shocks because of low or high impedance
CPR guidance initiated (i-button pushed) | Up to 15 minutes during device placement
  Percentage of events where CPR guidance was initiated (i-button pushed)
CPR activity | Up to 15 minutes during device placement
  Percentage of events where CPR is performed during CPR guidance

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit Noordergraaf, MD PhD, Principal Investigator — Philips Healthcare
Locations (1):
- Philips, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No